CLINICAL TRIAL: NCT01065051
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Study to Assess the Effects of a Single Dose of 1 mg Riociguat (BAY63-2521) on Myocardial Contractility and Relaxation in Patients With Pulmonary Hypertension Associated With Left Ventricular Systolic Dysfunction (PH-sLVD)
Brief Title: Hemodynamic and Echocardiographic Assessment of Riociguat Effects on Myocardial Wall Contractility and Relaxation Kinetics
Acronym: HEARTWORK
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14549
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension, Pulmonary; Ventricular Dysfunction, Left
Keywords: Pulmonary Hypertension; Left ventricular dysfunction
MeSH Terms: conditions — Hypertension, Pulmonary; Ventricular Dysfunction, Left | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Riociguat (Adempas, BAY63-2521) (Experimental): Participants received a single oral dose of 1 mg riociguat.
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)
- Placebo (Placebo Comparator): Participants received a single oral dose of 1 mg placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — 1 mg single oral dose
  Arms: Riociguat (Adempas, BAY63-2521)
Drug: Placebo — Single oral dose
  Arms: Placebo

SUMMARY:
The aim of this study is to assess whether oral Riociguat affects the left ventricular contractility and relaxation in patients with pulmonary hypertension associated with left ventricular systolic dysfunction

DETAILED DESCRIPTION:
Adverse event data will be covered in Adverse events section.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with symptomatic pulmonary hypertension due to left ventricular systolic dysfunction despite standard heart failure therapy

Exclusion Criteria:

* Types of pulmonary hypertension other than group 2.1 of Dana Point Classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Boston, Massachusetts
  - Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only subjects symptomatic with pulmonary hypertension associated with left ventricular systolic dysfunction (PH-sLVD) could participate in this study.
Pre-assignment Details: One subject was screened, randomized and treated during this study. The subject completed the study according to protocol.
Period: Overall Study
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Customized [Number; unit: Participants]
  <65 years | 0 |  | 0
  >=65 years | 1 |  | 1
Gender [Number; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Power Index at Rest
Description: The peak power index is a calculated hemodynamic parameter. It is derived from the directly measured parameters mean systolic arterial pressure (SAPmean) and mean pulmonary capillary wedge pressure (PCWPmean). These 2 parameters are acquired during a right heart catheterization. The peak power index is calculated from the maximal power (which also takes the calculated parameter cardiac output into account) divided by the left ventricular end-diastolic volume (LVEDV). Formula: Peak Power Index = (SAPmean - PCWPmean)*CO [cardiac output]*16.667/LVEDV
Time Frame: Before and 1 hour after administration of study drug
Population: Due to the very low number of patients enrolled in the study, no statistical evaluation was done.
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Left Ventricular Stroke Work Index (LVSWI) at Rest
Description: The left ventricular stroke work index (LVSWI) is a calculated hemodynamic parameter. It is derived from the directly measured parameters mean systolic arterial pressure (SAPmean) and mean pulmonary capillary wedge pressure (PCWPmean). These 2 parameters are acquired during a right heart catheterization. The LVSWI is also dependent of the calculated hemodynamic parameter stroke volume index (SVI). Formula: LVSWI = (SAPmean - PCWPmean)*SVI*0.0136
Time Frame: Before and 1 hour after administration of study drug
Population: Due to the very low number of patients enrolled in the study, no statistical evaluation was done.
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF) at Rest
Description: The left ventricular ejection fraction work index (LVEF) is a calculated echocardiography parameter. LVEF is derived from the directly measured parameters left ventricular end-diastolic volume (LVEDV) and left ventricular end-systolic volume (LVESV). These 2 parameters are acquired during a non-invasive echocardiography examination. Formula: LEVF = 100*(LVEDV - LVESV)/LVEDV
Time Frame: Before and 1 hour after administration of study drug
Population: Due to the very low number of patients enrolled in the study, no statistical evaluation was done.
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in End-systolic Elastance at Rest
Description: The end-systolic elastance is a calculated hemodynamic parameter. It is approximated by the directly measured hemodynamic parameter end-systolic pressure divided by the directly measured echocardiography parameter left ventricular end-systolic volume (LVESV). The end-systolic pressure is acquired during a right heart catheterization. The LVESV is acquired during a non-invasive echocardiography examination. Approximated by end-systolic pressure/LVESV
Time Frame: Before and 1 hour after administration of study drug
Population: Due to the very low number of patients enrolled in the study, no statistical evaluation was done.
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Peak Power Index During the Cardiopulmonary Exercise Tests
Description: The peak power index is a calculated hemodynamic parameter. It is derived from the directly measured parameters mean systolic arterial pressure (SAPmean) and mean pulmonary capillary wedge pressure (PCWPmean). These 2 parameters are acquired during a right heart catheterization. Formula: Peak Power Index = (SAPmean - PCWPmean)*CO*16.667/LVEDV
Time Frame: Before and 1 hour after administration of study drug
Population: Due to the very low number of patients enrolled in the study, no statistical evaluation was done.
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Lateral Mitral Annular Peak Systolic Velocity (Sm) During the Cardiopulmonary Exercise Tests
Description: The lateral mitral annular peak systolic velocity (Sm) is a measured echocardiography parameter. It is acquired during a non-invasive echocardiography examination.
Time Frame: Before and 1 hour after administration of study drug
Population: Due to the very low number of patients enrolled in the study, no statistical evaluation was done.
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Peak Systolic Tricuspid Annular Velocity (RV-Sm) During the Cardiopulmonary Exercise Tests
Description: The peak systolic tricuspid annular velocity (RV-Sm) is a measured echocardiography parameter. It is acquired during a non-invasive echocardiography examination.
Time Frame: Before and 1 hour after administration of study drug
Population: Due to the very low number of patients enrolled in the study, no statistical evaluation was done.
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Tricuspid Annular Plane Systolic Excursion (TAPSE) During the Cardiopulmonary Exercise Tests
Description: The tricuspid annular plane systolic excursion (TAPSE) is a measured echocardiography parameter. It is acquired during a non-invasive echocardiography examination.
Time Frame: Before and 1 hour after administration of study drug
Population: Due to the very low number of patients enrolled in the study, no statistical evaluation was done.
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Lateral Mitral Annular Peak Early Diastolic Velocity (E') During the Cardiopulmonary Exercise Tests
Description: The lateral mitral annular peak early diastolic velocity (E') is a measured echocardiography parameter. It is acquired during a non-invasive echocardiography examination.
Time Frame: Before and 1 hour after administration of study drug
Population: Due to the very low number of patients enrolled in the study, no statistical evaluation was done.
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in the Slope of the Relationship Between Work Rate and Mean Pulmonary Arterial Pressure (PAPmean) During the Cardiopulmonary Exercise Tests
Description: The slope of the relationship between work rate during cardiopulmonary exercise tests and PAPmean is derived from the directly measured hemodynamic parameter mean pulmonary arterial pressure (PAPmean). PAPmean is acquired during a right heart catheterization.
Time Frame: Before and 1 hour after administration of study drug
Population: Due to the very low number of patients enrolled in the study, no statistical evaluation was done.
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in the Ventilatory Efficiency (V'E/V'CO2) Measured From Baseline to the Anaerobic Threshold (AT) During the Cardiopulmonary Exercise Tests (CPET)
Description: Ventilatory efficiency (V'E/V'CO2) and anaerobic threshold (AT) were parameters directly measured or derived by computed analysis from the spiroergometry system during the cardiopulmonary exercise test.
Time Frame: Before and 1 hour after administration of study drug
Population: Due to the very low number of patients enrolled in the study, no statistical evaluation was done.
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to low recruitment (one subject enrolled only). No statistical analyses of efficacy parameters were performed. Therefore, no clinically meaningful conclusions can be drawn from the data generated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigative Site, Institution and/or Principal Investigator shall furnish the Sponsor with a copy of any proposed publication of material described in Clinical Trial Agreement at least sixty (60) days in advance of the date of submission for publication or presentation. Within sixty (60) day period, the Sponsor shall: review such proposed publication for any patentable subject matter or designated Confidential Information, which the Sponsor may have furnished to facilitate the study.